CLINICAL TRIAL: NCT03832439
Title: The Effect of Probiotic Supplementation on Weight Loss, and Its Association With the Gut Microbiome After Bariatric Surgery.
Brief Title: Probiotic Supplementation on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Meera Shah, M.B., Ch.B., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-003300
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Bariatric Surgery Candidate
Keywords: Probiotic; Microbiome
MeSH Terms: interventions — Probiotics; microcrystalline cellulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): This arm will be receiving probiotic supplements.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): This arm will be receiving placebo containing microcrystalline cellulose.
  Interventions: Dietary Supplement: microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: Probiotic — Lactobacillus rhamnosus GG 10 billion cells and microcrystalline cellulose
  Other Names: Culturelle®
  Arms: Probiotic
Dietary Supplement: microcrystalline cellulose — Placebo
  Arms: Placebo

SUMMARY:
The investigators are trying to better understand how bariatric surgery leads to weight loss, and the role of bacteria that live in the gut in making this happen.

DETAILED DESCRIPTION:
The investigators are interested in seeing how a probiotic, which is a dietary supplement containing large amounts of 'good' bacteria, can influence the make-up of the gut bacterial population and what effect it has on weight loss and loss of fat. Before undergoing weight loss surgery (sleeve gastrectomy or roux-en-y gastric bypass), study participants will be asked to provide a stool sample to assess the make-up of their gut bacterial population. They will also undergo a limited CT scan of the abdomen and DEXA (Xray) to help assess the amount of fat present inside the body.

After undergoing weight loss surgery (sleeve gastrectomy or roux-en-y gastric bypass), study participants will be given either a probiotic supplement or dummy pill (placebo) for 3 months, in addition to all usual care that occurs after surgery. The CT scan, DEXA scan and stool sample will be repeated at the end of the 3 month period and analyzed for changes.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects who are > 18 and < 65 years of age recruited from the Mayo Clinic bariatric surgery clinic
2. Will also meet one of the National Institute of Health's criteria for bariatric surgery, i.e. body mass index (BMI) > 40 kg/m2 or BMI > 35 kg/m2 with significant weight-related comorbidities.
3. Patients will be eligible if they are not on chronic antibiotic therapy and without active systemic illness.

Exclusion Criteria:

1. Patients with type 1 or 2 diabetes will be excluded due to the known pre-existing changes in the gut microbiome in this population. All patients will not have had exposure to probiotics, prebiotics or antibiotics in the preceding 4 weeks.
2. Patients with allergy to antibiotics precluding the use of standard peri-operative antibiotics (cefazolin and metronidazole) will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Weight loss | 3 months
  Change in body weight from baseline to 3 months
Visceral fat loss | 3 months
  Change in visceral fat from baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Meera Shah, M.B., Ch.B, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials